CLINICAL TRIAL: NCT02347540
Title: Queen of Hearts Research Program. Identifying the Risk on Heart Failure After Preeclampsia.
Brief Title: Heart Failure and Related Risk-factors After Preeclampsia
Acronym: QoH
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University Medical Center (Other)
Collaborators: UMC Utrecht (Other); Leiden University Medical Center (Other); University Medical Center Groningen (Other); Amsterdam UMC, location VUmc (Other); Dutch Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: METC 14-02-013; 2013T084 (Other Grant/Funding Number: Nederlandse Hartstichting (Dutch Heart Foundation))
Record Dates: First submitted 2014-12-30; First posted 2015-01-27 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Heart Failure; Cardiovascular Diseases; Pre-Eclampsia
Keywords: Heart Failure; Diastolic Dysfunction; Pre-Eclampsia; Endothelial dysfunction; Biological Markers; MicroRNAs; Circulating cells
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators will perform an unbiased screen for the human genome content of circulating microRNAs. HF biomarkers will be included so that the added value of these novel HFpEF miRNAs can directly be compared to established HF biomarkers. In this cohort of women who experienced pre-eclampsia and matched controls, the investigators will profile miRNAs on a genome-wide scale using total RNA from plasma. Differentially expressed miRNAs will be further investigated in relation to the pathogenesis of micro- and macrovascular disease. Selected miRNAs will be placed on a custom megaplex array and used to screen a cohort of patients with HFpEF. In patients with HFpEF the investigators will relate miRNA expression level to the circulating levels of angiopoietin-2/ang-1ratio's and micro-albuminuria. Part of the obtained blood and urine will be stored at the Biobank in Maastricht for future studies.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Women with a history of preeclampsia (cases): Cases: women with a history of preeclampsia. Measurements will be performed in a postpartum interval from 0.5 years until 30 years after the first complicated pregnancy.
  This group will further be subdivided in a subgroup with Heart Failure and a group without Heart Failure.
- Women with a history of uncomplicated pregnancy (controls): Controls include women with a history of uncomplicated pregnancies. The controlgroup will further be subdivided in a subgroup with Heart Failure and a group without Heart Failure.

SUMMARY:
This study is a cross-sectional case-control study where classical as well as more innovative risk factors for CVD will be explored.

In western countries, more women than men die of cardiovascular disease (CVD), making CVD in women an important public health issue. Misdiagnosis of CVD in women is frequently observed, posing the clinician for diagnostic and therapeutic dilemmas that can easily result in inadequate treatment and worse prognosis. Despite these challenges, CVD in women has been underexposed in scientific research.

Women have gender-specific risk factors like a history of preeclampsia (PE) that contribute to their risk for CVD. PE complicates 5-10% of pregnancies, recurs in ~25% and is associated with a 2-4 fold increased risk for CVD. Moreover, pre-symptomatic heart failure (HF) stage B occurs in 40% of women with a history of PE. HF stage B is thought to precede the development of the, mortality related, clinical HF stages C and D (structural heart disease in combination with symptomatic disease). Early detection and tailored intervention of women with stage B HF decreases progression to the clinical stages and might therefore improve clinical outcome and cardiovascular related mortality.

Phenotypic presentation of HF is currently split up between systolic HF also called HF with reduced ejection fraction (HFrEF) and diastolic HF or HF with preserved ejection fraction (HFpEF). Women more often have HFpEF in contrast to men. Different pathophysiology and disease progression in women compared to men seems to be an important underlying factor. The current clinical HF diagnostic tools (e.g. natriuretic hormones and high sensitivity troponins) fail to identify early changes that prelude adverse cardiac remodelling and HF, and do not discriminate between HFrEF and HFpEF. Moreover, there are sex-related differences in biomarker levels for detection of CVD. As a result, clinicians are forced to wait for the failing heart to become clinically evident before they can intervene. Therefore, there is an urgent need to assess novel biomarkers that could help select high risk women needing further follow up and intervention. Biomarkers may not only improve early diagnosis but may also unravel disease pathways of HFpEF. Especially when combined with measurements of subclinical, surrogate risk markers.

Objectives

* To determine the impact of PE on incidence of macro-and micro-vascular dysfunction reflected by surrogate measures for coronary artery disease (CAD) and HFpEF.
* To perform a genome wide association study (GWAS) and associate novel biomarker expression levels with endothelial function, cardiac diastolic function and IMT measurement.
* To identify risk factors and surrogate measures for CVD in a) former PE patients without HFpEF, b) former PE patients with HFpEF and c) healthy parous controls.

Study population Cases: women with a history of PE Controls: women with uncomplicated pregnancies in the history. Measurements will be performed in clusters at postpartum intervals of: ½-2, 5-10, 10-15 and 15-30 years. Number of inclusions will be: 425, 350, 282 and 233 for each follow-up group respectively.

Primary endpoints The prevalence of macro- and microvascular dysfunction in former PE patients. Novel biomarker detection in former PE patients associated with HF in general and HFpEF in particular.

Secondary endpoints

* Lifestyle (questionnaire)
* Cognitive ability (questionnaire)
* Depression score (questionnaire)
* Metabolic syndrome (MetS)
* Arterial endothelial function (Flow mediated dilation (FMD))
* Intima Media Thickness (IMT)
* Glycocalyx thickness (by means of the Glycocheck)
* Venous function (plethysmograph)
* Electrocardiogram (ECG)
* Ergometry

ELIGIBILITY:
Inclusion Criteria:

Cases

* Women aged ≥ 18 years
* ½ till 30 years after the complicated pregnancy
* Experienced PE in any pregnancy. PE defined as hypertension (systolic BP ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg) developed after 20 weeks of pregnancy with the development of proteinuria (≥ 300 mg/ 24 hours).
* Women who had their last delivery at least 6 months ago.

Controls

* Women aged ≥ 18 years
* ½ till 30 years after the pregnancy that matches the sequence number of pregnancy of the specifically matched case.
* Experienced pregnancies that were not complicated by foetal or maternal placental syndrome (pregnancy induced hypertension, preeclampsia, HELLP-syndrome).
* Women who had their last pregnancy at least 6 months ago.
* Women with a negative family history for PE (mother and sisters did not experience PE).

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

Cases

* Women with auto-immune diseases prior to the complicated pregnancy.
* Chronic hypertension prior to the complicated pregnancy.
* Renal disease prior to the complicated pregnancy.
* Pregnant women
* Women who do not want to be informed about the results of the tests, or women who do not want their general practitioner and specialist(s) to be informed about the test results.

Control group:

* Women with auto-immune diseases
* Chronic hypertension prior to the matched pregnancy.
* Women with IUGR in the matching pregnancy (p<10)
* Solutio placentae in the matching pregnancy
* Pregnant women
* Women who do not want to be informed about the results of the tests, or women who do not want their general practitioner and specialist(s) to be informed about the test results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: women with a history of PE. Control group: women with uncomplicated pregnancies in the history H1: PP interval ½ -2 years: n = 2x 425 H2: PP interval 5-10 years: n = 2x 350 H3: PP interval 10-15 years: n = 2x 282 H4: PP interval 15-30 years: n = 2x 233
Sampling Method: Probability Sample
Enrollment: 2580 (Estimated)
Dates: Start 2014-12 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The prevalence of Heart Failure (number with percentage) | At time of assessment
  Heart Failure will be assessed with the transthoracic echocardiography based on the criteria of the American Heart Association. The sub classification for Heart Failure with preserved ejection fraction (EF) will be made (EF >55%)

SECONDARY OUTCOMES:
Structural en Functional Cardiac Measurements | At time of assessment
  The objective is to estimate structural and functional cardiac measurements with the TTE based on the ASA guidelines.
Metabolic syndrome | At time of assessment
  The objective is to assess the prevalence of constituents of the Metabolic syndrome based on the WHO criteria. The prevalence will be reported in number with percentage.
Arterial endothelial function (Flow mediated dilation (FMD)) | At time of assessment
  The objective is to estimate NO mediated endothelial function of the brachial artery with ultrasound by FMD and sublingual NTG administration. FMD will be reported in relative increase in diameter (%).
Common Carotid Intima media thickness | At time of assessment
  The objective is to estimate IMT of the common carotid artery in cm using ultrasound.
Glycocalyx thickness en microvascular tortuosity | At time of assessment
  The objective is to estimate the glycocalyx dimensions using sublingual orthogonal polarization spectral (OPS) measurements. Derivative of the glycocalyx (perfused boundary region) will be reported in um. Tortuosity will be reported based on a score system.
Cognitive, Lifestyle and Depression rates | At time of assessment
  To evaluate subjective cognitive functioning and depression rates and lifestyle behavior in formerly preeclamptic women with heart failure compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Marc EA Spaanderman, MD, PhD, Study Chair — Maastricht University Medical Center; Gerard Pasterkamp, PhD, Study Chair — UMC Utrecht; Hester HM den Ruijter, PhD, Study Chair — UMC Utrecht
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Brandt Y, Alers RJ, Canjels LPW, Jorissen LM, Jansen G, Janssen EBNJ, van Kuijk S, Went TM, Koehn D, Gerretsen SC, Jansen J, Backes W, Hurks PPM, van de Ven V, Kooi ME, Spaanderman MEA, Ghossein-Doha C. DEcreased Cognitive functiON, NEurovascular CorrelaTes and myocardial changes in women with a history of pre-eclampsia (DECONNECT): research protocol for a cross-sectional pilot study. BMJ Open. 2024 Mar 4;14(3):e077534. doi: 10.1136/bmjopen-2023-077534. PMID 38443087
- [Derived] Mohseni-Alsalhi Z, B N J Janssen E, Delmarque J, van Kuijk SMJ, Spaanderman MEA, Ghossein-Doha C. Prediction Model Based on Easily Available Markers for Aberrant Cardiac Remodeling in Women After Pregnancy. Hypertension. 2023 Aug;80(8):1707-1715. doi: 10.1161/HYPERTENSIONAHA.122.19187. Epub 2023 Jan 25. PMID 37470772
- [Derived] Alers RJ, Ghossein-Doha C, Canjels LPW, Muijtjens ESH, Brandt Y, Kooi ME, Gerretsen SC, Jansen JFA, Backes WH, Hurks PPM, van de Ven V, Spaanderman MEA. Attenuated cognitive functioning decades after preeclampsia. Am J Obstet Gynecol. 2023 Sep;229(3):294.e1-294.e14. doi: 10.1016/j.ajog.2023.02.020. Epub 2023 Feb 28. PMID 36863645
- [Derived] Janssen EBNJ, Hooijschuur MCE, Lopes van Balen VA, Morina-Shijaku E, Spaan JJ, Mulder EG, Hoeks AP, Reesink KD, van Kuijk SMJ, Van't Hof A, van Bussel BCT, Spaanderman MEA, Ghossein-Doha C. No accelerated arterial aging in relatively young women after preeclampsia as compared to normotensive pregnancy. Front Cardiovasc Med. 2022 Jul 28;9:911603. doi: 10.3389/fcvm.2022.911603. eCollection 2022. PMID 35966519